CLINICAL TRIAL: NCT03680378
Title: A Phase I Open-Label, Single-Centre Study to Assess the Concentration of AAI101 and Cefepime in Epithelial Lining Fluid and Plasma in Healthy Volunteers
Brief Title: Lung Pharmacokinetics (PK) in Epithelial Lining Fluid (ELF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allecra (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AT-103
Record Dates: First submitted 2018-07-25; First posted 2018-09-21 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Healthy Subjects
Keywords: bronchial epithelial lining fluid
MeSH Terms: interventions — enmetazobactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cefepime 2 gram + AAI101 1 gram (Experimental): cefepime 2 grams in combination with AAI101 1 gram intravenous infusion
  Interventions: Drug: Cefepime 2 gram

INTERVENTIONS:
Drug: Cefepime 2 gram — Combination of cefepime 2 gram with AAI101 1 gram
  Other Names: AAI101

SUMMARY:
The primary objective of this study is to measure and compare the concentration of AAI101 and cefepime in bronchial epithelial lining fluid (ELF) and plasma following administration of cefepime/AAI101 combination in healthy subjects.

ELIGIBILITY:
1. Provision of signed and dated, written informed consent prior to any study-specific procedures.
2. Healthy male and female subjects aged 18 to 65 years with veins suitable for cannulation or repeated venipuncture. Female patients can participate if at least 1 of the following criteria are met:

   * Are of non-childbearing potential defined as
   * Permanently sterile following hysterectomy, bilateral salpingectomy, bilateral oophorectomy or confirmed tubal occlusion (not tubal ligation);
   * Postmenopausal, as defined as at least 1 year post-cessation of menses (without an alternative medical cause), and per documentation provided by a medical professional;
   * Postmenopausal status will be confirmed with a screening serum follicle stimulating hormone (FSH) level greater than 40 milli-international units per milliliter (mlU/mL).
   * Patient has a negative urine and/or serum pregnancy test (serum β-human chorionic gonadotropin) within 1 day prior to study entry, and agrees to use highly effective contraception methods during treatment and for at least 7 days after the last dose of i.v. study therapy;
3. Have a body mass index (BMI) between 18 and 32 kg/m2.
4. As judged by the Investigator, all the subjects must be able to understand and be willing to comply with study procedures, restrictions and requirements.

4.2 Exclusion criteria

Subjects should not enter the study if any of the following exclusion criteria are fulfilled:

1. Male subjects who do not agree to follow contraception restrictions.
2. Female subjects who are pregnant or currently lactating
3. Female subjects who are of child bearing potential who do not agree to follow contraception restrictions as detailed in section 5.1.10.
4. Donated blood in the 3 months prior to screening, plasma in the 7 days prior to screening, platelets in the 6 weeks prior to screening
5. Consume more than 28 units of alcohol per week if male, or 21 units of alcohol per week if female or any significant history of alcohol / substance misuse as determined by the investigator
6. Unwilling to abstain from vigorous exercise for 48 hours prior to any study visit
7. Unwilling to abstain from alcohol for 48 hours prior to any study visit
8. Used cigarettes or vapor e-cigarettes, cigars or other nicotine-containing products (with the exception of nicotine replacement products not covered above) within 3 months before bronchoscopy or have a smoking history greater than 10 pack years.
9. Received any medication, including St John's Wort, known to chronically alter drug absorption or elimination within 30 days prior to first dose administration unless in the opinion of the investigator it will not interfere with study procedures or compromise safety
10. Received any prescribed systemic or topical medication within 14 days prior to the first dose administration (with the exception of the oral contraceptive pill)
11. Received any non-prescribed systemic or topical medication, herbal remedy or vitamin / mineral supplementation within 14 days prior to the first dose administration (with the exception of paracetamol).
12. Subjects who have any abnormality of vital signs prior to the first dose administration that, in the opinion of the investigator, would increase the risk of participating in the study
13. Subjects who have any clinically significant abnormal physical examination finding
14. Subjects who have any clinically significant 12 lead ECG abnormality that, in the opinion of the investigator, would increase the risk of participating in the study
15. Subjects who have, or have any history of, any clinically significant cardiovascular, respiratory, gastrointestinal, neurological, psychiatric, metabolic, endocrine, renal, hepatic, haematological or other major disorder as determined by the investigator
16. Subjects who have any significant condition that may preclude nasal or oral intubation with a bronchoscope as determined by the investigator
17. Subjects who have any clinically significant allergy or allergic condition as determined by the investigator (with the exception of non-active hay fever)
18. Subjects who have had previous adverse reactions to benzodiazepines or anaesthetic agents (lidocaine or xylocaine) including reversal agents such as flumazenil
19. Subjects who have any clinically significant abnormal laboratory safety results as determined by the investigator with specific exclusions of any aspartate aminotransferase (AST) or alanine aminotransferase (ALT)upper limit of normal greater than or equal to 1.5 times upper limit of normal (ULN) at screening or day -1; total bilirubin > ULN (Gilbert's syndrome is acceptable), haemoglobin <12.0 g/dL or prothrombin time > 13 seconds (one repeat assessment is acceptable at screening)
20. Subjects who have hepatitis B or C or are carriers of HBsAg or are carriers of hepatitis C virus (HCV= Ab or are positive for HIV 1/2 antibodies.
21. Subjects who have a positive alcohol breath test or a positive urine drug screen ( a repeat assessment is acceptable)
22. Subjects who are still participating in another clinical study or who have participated in a clinical study involving administration of an investigational product in the 3 months (or 5 half-lives, whichever is longer) prior to first dose administration
23. Subjects who, in the opinion of the investigator, should not participate in this study For procedures for withdrawal of incorrectly enrolled subjects, see Section 5.3. Subjects who drop out will be replaced.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of cefepime and AAI101 in the lung | Change from baseline to 2 hours, 4 hours, 6 hours and 8 hours post dose
  Maximum concentration of cefepime and AAI101 in Bronchoalveolar lavage (BAL) samples

SECONDARY OUTCOMES:
Maximum concentration of cefepime and AAI101 in plasma | Change from baseline to 2 hours, 4 hours, 6 hours and 8 hours post dose
  Maximum concentration of cefepime and AAI101 in plasma samples

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No